CLINICAL TRIAL: NCT06743230
Title: The Effect of Neuroathletic Training on Physical Performance and Position Sense in Cross-country Skiers
Brief Title: The Effect of Neuroathletic Training in Cross-country Skiers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Nurcan Contarli, Lecturer, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KarabukUniv-FTR
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Skiing/Snowboarding
Keywords: Cross-Country Skiing; Neuroathletic Training; Strength; Balance; Proprioception

STUDY DESIGN:
Intervention Model Description: Two groups with a neuro athletic training group and a control group.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessments will be performed by an investigator who was blinded to group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Training (Active Comparator): Conventional training includes flexibility exercises, strengthening exercises, running, balance and sport-specific technique work 5 days per week.
  Interventions: Other: Conventional training
- Neuro athletic training (Experimental): Conventional training includes flexibility exercises, strengthening exercises, running, balance, and sport-specific technique work 5 days per week.Neuro athletic training includes exercises that stimulate the visual, vestibular and proprioceptive systems. The neuroathletic training includes 3 days per week for 8 weeks.
  Interventions: Other: Neuro athletic training; Other: Conventional training

INTERVENTIONS:
Other: Neuro athletic training — The neuroathletic training includes exercises that stimulate the visual, vestibular, and proprioceptive systems. The neuroathletic training includes 3 days per week for 8 weeks.
  Arms: Neuro athletic training
Other: Conventional training — Conventional training includes flexibility exercises, strengthening exercises, running, balance and sport-specific technique work 5 days per week.

SUMMARY:
The aim of this study was to investigate the effects of neuro-athletic training on physical performance and position sense in cross-country skiers.

DETAILED DESCRIPTION:
Cross-country skiing is the least dangerous but tiring winter sport performed in snowy environments with different heights, distances, and slopes using ski equipment such as skis, shoes, and poles with various features. In this sport, both the lower and upper body require rapid power production and high maximal oxygen consumption. When technique, conditioning, and skill are combined in cross-country skiing, the resulting performance reaches the highest level. In order for an athlete to perform well, they must have the capacity to produce power continuously and quickly. Cross-country skiing is often associated with the development of strength, speed, agility, balance, endurance, fatigue resistance, and oxygen capacity. Physical training alone is not enough for an athlete to achieve high success. Physical training must be combined with the visual system, vestibular system, and proprioceptive system. The quality of the stimuli coming from these systems in an athlete positively affects the athlete's physical performance and success in competitions. Therefore, in addition to the physical training that the athlete will do, neuro-athletic training that stimulates the visual, vestibular, and proprioceptive systems will be implemented in the cross-country skiing sports branch, considering that it can increase the athlete's performance by improving muscle strength, core endurance, balance, and proprioceptive sense. The sample of the study will consist of 26 cross-country skiing athletes between the ages of 12-18 who participate in training at the Arkut Cross-Country and Biathlon Center. The athletes will be randomly divided into 2 groups by coin toss method. All athletes will participate in routine training. Neuroathletic training will be given to one group in addition to routine training, and its effect on the athletes' performance will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Have been cross-country skiing for at least 3 years and regularly participate in training
* Be a volunteer
* Complete a Trail Making Test

Exclusion Criteria:

* Have had lower extremity surgery in the last 2 years
* Have no neurological or orthopedic disorders

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Knee Joint Position Sense | 8 weeks
  Knee joint position sense will be measured using the passive-active repositioning method with a digital inclinometer.
Dynamic balance | 8 weeks
  Dynamic balance will be evaluated with the Y balance test.
Muscle strength | 8 weeks
  Knee flexion and extension isometric muscle strength will be measured with a handheld dynamometer.
Trunk Flexion Endurance Test | 8 weeks
  The time that athletes can maintain a stance with their trunk at 60° flexion and their hips and knees at 90° flexion will be measured with a stopwatch.
Side Bridge Endurance Test | 8 weeks
  Athletes will be asked to perform a side bridge in a side-lying position, with legs extended, one foot in front of the other, the body in a straight line, with the elbow joint flexed on the same side, supported by the forearm. The time they can maintain this position will be recorded with a stopwatch.
Slalom Test | 8 weeks
  For this test, 6 cones will be placed on a 12-meter track at 2-meter intervals. Athletes were asked to run between the cones at maximum speed and the elapsed time will be recorded with a stopwatch.

CONTACTS AND LOCATIONS:
Overall Officials: Necmiye UnYildirim Professor, PhD, Study Director — Saglik Bilimleri Universitesi; Caglar Soylu Assistant Professor, PhD, Study Director — Saglik Bilimleri Universitesi
Locations (1):
- Arkut Cross-Country Skiing and Biathlon Center, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No